CLINICAL TRIAL: NCT06343051
Title: Ultrasound Hemodynamic Assessment in Newly Diagnosed Fetal Growth Restriction: A Pilot Study
Brief Title: USCOM in Newly Diagnosed FGR Cases
Acronym: USCOM FGR
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Rachel Meislin, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-23-01681
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-07

CONDITIONS: Fetal Growth Restriction; USCOM
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Fetal Growth Restriction diagnosed > 27w6d gestation: Patients with a new diagnosis of fetal growth restriction after 27 weeks 6 days' gestation.
  Interventions: Device: USCOM

INTERVENTIONS:
Device: USCOM — Device that measures how much blood is being pumped in and out of the heart.

SUMMARY:
The purpose of this research study is to study the use of an ultrasound measurement system (USCOM) for patients with newly diagnosed fetal growth restriction (FGR). This system uses a technology to measure how much blood is being pumped in and out of the heart, which is important for understanding the heart's function in relation to pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with a new diagnosis of fetal growth restriction (estimated fetal weight <10th percentile or abdominal circumference <10th percentile) in the third trimester (gestational age >27w6d)

Exclusion Criteria:

* Multiple gestation
* Fetal anomalies
* Gestational diabetes or pregestational diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed fetal growth restriction at greater than 27 weeks 6 days' gestation will be eligible to enroll in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Systemic vascular resistance obtained from USCOM | every 2-4 weeks at time of prenatal ultrasound, until the end of pregnancy
  Cardiac output related to systemic vascular resistance (SVR) obtained from the USCOM device. SVR is an indicator of general resistance experienced within the circulatory system and is correlated with an array of cardiac related adverse health outcomes. The USCOM device uses noninvasive ultrasonographic technology to determine SVR at the time of prenatal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola F Tavella, MPH, Study Director — Icahn School of Medicine at Mount Sinai; Rachel J Meislin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to Nicola.tavella@mssm.edu. To gain access, data requestors will need to sign a data access agreement.